CLINICAL TRIAL: NCT00257595
Title: Long-term Study of Cetirizine Dry Syrup in Children. Suffering From Perennial Allergic Rhinitis.
Brief Title: Perennial Allergic Rhinitis In Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104914
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial Allergic Rhinitis pediatric
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetirizine Dry Syrup

SUMMARY:
To assess the safety of long-term use of cetirizine dry syrup in children with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Children with perennial allergic rhinitis.
* Giving informed consent.
* Children with a positive response to specific IgE antibody test.
* Children assessed as positive in the nasal eosinophil count.
* Children whose severity score of nasal symptom is 4 or higher.

Exclusion criteria:

* have a history of drug hypersensitivity.
* are pregnant, lactating or possibly pregnant female children.
* Sensitivity to pollen as a duplicate allergen and whose treatment periods are thought in the pollen dispersion periods.
* have vasomotor rhinitis and eosinophilic rhinitis.
* have asthma that requires the treatment with corticosteroid.
* have inappropriate complication of nasal disorder that may influence on the evaluation of the study drugs.
* have complicated with atopic dermatitis or urticaria that requires the treatment with antihistamine preparation.
* have started specific desensitization treatment.
* nonspecific modulation treatment but who have not reached the maintenance level of treatment.
* have received surgical treatment for reduction and modulation of nasal mucosa.
* redintegration therapy of nasal cavity to improve the degree of nasal airway.
* surgical operation to improve rhinorrhea.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2005-08

PRIMARY OUTCOMES:
safety

SECONDARY OUTCOMES:
Total Nasal Symptom Score (TNSS) Individual nasal symptom score total score of 4 individual daily symptom scores Investigator global improvement rating

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site